CLINICAL TRIAL: NCT04767451
Title: Levels of Selected Microelements in Premature Ovarian Insufficiency
Acronym: POI&MICROs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cengiz Gokcek Women's and Children's Hospital (Other)
Responsible Party: Principal Investigator, Ali Ovayolu, Principal Investigator, Cengiz Gokcek Women's and Children's Hospital
Other Study IDs: CengizGWCH22
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Premature Ovarian Failure
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Premature ovarian insufficiency (POI): POI is a clinical syndrome defined by loss of ovarian activity before the age of 40 years. POI is characterized by menstrual disturbance (amenorrhea or oligomenorrhea) with raised gonadotropins and low estradiol.
  Interventions: Diagnostic Test: ultrasound assessment
- Control group: The study population will consist of 50 women with POI as a study group and 50 patients with normal healthy women as a control group. A volunteer group of healthy women who will be visited the gynecology clinic for routine examinations and women who will be admitted for pre-pregnancy tests will be invited randomly to this research as a control group.
  Interventions: Diagnostic Test: ultrasound assessment

INTERVENTIONS:
Diagnostic Test: ultrasound assessment — Lead (Pb), Cadmium (Cd), Gadolinium (Gd), Arsenic (As), Mercury (Hg), Cobalt (Co), Vanadium (V), Titanium (Ti), Sulfur (S), Chromium (Cr), Silver (Ag), Molybdenum (Mo), Boron (B), Lithium (Li), and Nickel (Ni) measurements

SUMMARY:
Aim: To evaluate plasma/urine/hair Lead (Pb), Cadmium (Cd), Gadolinium (Gd), Arsenic (As), Mercury (Hg), Cobalt (Co), Vanadium (V), Titanium (Ti), Sulfur (S), Chromium (Cr), Silver (Ag), Molybdenum (Mo), Boron (B), Lithium (Li), and Nickel (Ni) levels in women with premature ovarian insufficiency (POI) and to compare the results with those of healthy subjects.

Methods: This prospective study will be included 50 women with idiopathic premature ovarian insufficiency and 50 controls. The blood/urine/hair for analyses will be obtained at the early follicular phase of the menstrual cycle and plasma Lead (Pb), Cadmium (Cd), Gadolinium (Gd), Arsenic (As), Mercury (Hg), Cobalt (Co), Vanadium (V), Titanium (Ti), Sulfur (S), Chromium (Cr), Silver (Ag), Molybdenum (Mo), Boron (B), Lithium (Li), and Nickel (Ni) levels will be measured using inductively coupled plasma-mass spectrometry.

DETAILED DESCRIPTION:
This will be an observational prospective cohort study conducted at Obstetrics and Gynecology Department of Cengiz Gokcek Obstetrics and Children's Hospital between January 2020 and June 2021. The authors will be recruited 50 subjects with idiopathic POI, and 50 healthy patients were selected for the control group. All patients will be given their oral and written informed consent before their inclusion in the study. The protocol was approved by the Ethics Committee for Clinical Research of Gaziantep University (Reference number: 2020/320). The study strictly will be adhered to the principles of the Declaration of Helsinki.

Women between the ages of 18-39 will be included. A volunteer group of healthy women who will be visited the gynecology clinic for routine examinations and women who will be admitted for pre-pregnancy tests will be invited randomly to this research as a control group. Healthy women, who will be returned during their early follicular phase of the menstrual cycle, will be recruited as the control group subjects. The exclusion criteria will be as follows: women with evidence for karyotypic, metabolic, toxic, or iatrogenic cause of the ovarian insufficiency and any women who use any medication for POI treatment. At enrollment, for both groups, the authors will be collected data about age, height, weight, BMI, age of menarche, obstetrics history, history of smoking, regular exercise and family history of POI. At enrolment, all patients will be underwent vaginal ultrasonography for the assessment of antral follicle count (AFC) and venous blood sample from the antecubital veins for measuring plasma concentration of Lead (Pb), Cadmium (Cd), Gadolinium (Gd), Arsenic (As), Mercury (Hg), Cobalt (Co), Vanadium (V), Titanium (Ti), Sulfur (S), Chromium (Cr), Silver (Ag), Molybdenum (Mo), Boron (B), Lithium (Li), and Nickel (Ni), Follicle-stimulating hormone (FSH), E2, anti-mullerian hormone (AMH) and complete blood count (CBC). In control subjects venous blood samples and AFC will be collected during the early follicular phase of the menstrual cycle. Urine and hair samples will be collected at the same time. The plasma and urine samples will be stored in aliquots at -80°C prior to the analyses of Lead (Pb), Cadmium (Cd), Gadolinium (Gd), Arsenic (As), Mercury (Hg), Cobalt (Co), Vanadium (V), Titanium (Ti), Sulfur (S), Chromium (Cr), Silver (Ag), Molybdenum (Mo), Boron (B), Lithium (Li), and Nickel (Ni). Hair samples will be stored in envelopes at room temperature. The plasma/urine/hair Lead (Pb), Cadmium (Cd), Gadolinium (Gd), Arsenic (As), Mercury (Hg), Cobalt (Co), Vanadium (V), Titanium (Ti), Sulfur (S), Chromium (Cr), Silver (Ag), Molybdenum (Mo), Boron (B), Lithium (Li), and Nickel (Ni) level will be measured using inductively coupled plasma-mass spectrometry. Then, this study will be determined plasma/urine/hair Lead (Pb), Cadmium (Cd), Gadolinium (Gd), Arsenic (As), Mercury (Hg), Cobalt (Co), Vanadium (V), Titanium (Ti), Sulfur (S), Chromium (Cr), Silver (Ag), Molybdenum (Mo), Boron (B), Lithium (Li), and Nickel (Ni) levels in women with POI (n=50) compared to those of volunteer healthy women (n=50). Then, these microelements levels will be compared in both group.

ELIGIBILITY:
Inclusion Criteria:

* women with idiopathic POI
* Healthy women

Exclusion Criteria:

1. women with any systemic condition (such as chronic hypertension, renal disease)
2. history of using any medication
3. drug user
4. history/presence of malignancy
5. history of Radiotherapy/chemotherapy
6. polycystic ovary syndrome
7. endometriosis
8. Patients whose chromosome analysis result is not normal
9. history of ovarian surgery
10. Ovarian cysts/mass
11. pregnancy
12. lactation
13. women who get their hair coloured

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — POI is a clinical syndrome defined by loss of ovarian activity before the age of 40 years. POI is characterized by menstrual disturbance (amenorrhea or oligomenorrhea) with raised gonadotropins and low estradiol. It is estimated to affect 1% of women under the age of 40, 0.1% under 30 and 0.01% under 20.
Study Population: The investigators consecutively will be recruited 50 subjects with POI, and 50 healthy women will be selected for the control group.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Levels of selected microelements in POI | 1 week
  The primary outcome in these analyses will compare Lead (Pb), Cadmium (Cd), Gadolinium (Gd), Arsenic (As), Mercury (Hg), Cobalt (Co), Vanadium (V), Titanium (Ti), Sulfur (S), Chromium (Cr), Silver (Ag), Molybdenum (Mo), Boron (B), Lithium (Li), and Nickel (Ni) levels (µg/L,mean±SD) in the idiopathic POI group and control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Cengiz Gokcek Women's and Child's hospital, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] European Society for Human Reproduction and Embryology (ESHRE) Guideline Group on POI; Webber L, Davies M, Anderson R, Bartlett J, Braat D, Cartwright B, Cifkova R, de Muinck Keizer-Schrama S, Hogervorst E, Janse F, Liao L, Vlaisavljevic V, Zillikens C, Vermeulen N. ESHRE Guideline: management of women with premature ovarian insufficiency. Hum Reprod. 2016 May;31(5):926-37. doi: 10.1093/humrep/dew027. Epub 2016 Mar 22. PMID 27008889
- [Result] Pan W, Ye X, Zhu Z, Li C, Zhou J, Liu J. A case-control study of arsenic exposure with the risk of primary ovarian insufficiency in women. Environ Sci Pollut Res Int. 2020 Jul;27(20):25220-25229. doi: 10.1007/s11356-020-08806-0. Epub 2020 Apr 28. PMID 32347494
- [Result] Maclaran K, Horner E, Panay N. Premature ovarian failure: long-term sequelae. Menopause Int. 2010 Mar;16(1):38-41. doi: 10.1258/mi.2010.010014. No abstract available. PMID 20424285

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/51/NCT04767451/Prot_SAP_000.pdf